CLINICAL TRIAL: NCT04055454
Title: A Randomized, Placebo-controlled Trial to Evaluate the Optimal Dose of MV-LASV, a New Vaccine Against LASSA Virus Infection, Regarding Safety, Tolerability & Immunogenicity in Healthy Volunteers Consisting of an Unblinded Dose Escalation & an Observer-blinded Treatment Phase
Brief Title: A Trial to Evaluate the Optimal Dose of MV-LASV (V182-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Themis Bioscience GmbH (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other); Harmony Clinical Research BVBA (Other); Assign Data Management and Biostatistics GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V182-001; MV-LASV-101 (Other: Themisbio); 2018-003647-40 (EudraCT Number)
Record Dates: First submitted 2019-07-29; First posted 2019-08-13 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Lassa Virus Infection
Keywords: Lassa Virus Infection; Prevention; Vaccine; Phase 1; Lassa Fever
MeSH Terms: conditions — Lassa Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As safety precaution, the study will begin with enrollment of two successive unblinded dose groups of sentinel participants randomized into groups of four in an open-label fashion (group A and B). All site personnel, Sponsor and participants will be unblinded.
  Then remaining participants will be randomized in a blinded manner to one of three Treatment Groups (A, B, C). Site personnel responsible for study medication handling, preparation and Administration will be unblinded, only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MV-LASV low dose: treatment group A (Experimental): In total 24 participants will receive two low dose treatments with MV-LASV on day 0 and 28.
  Interventions: Biological: MV-LASV; Other: Placebo
- MV-LASV high dose: treatment group B (Experimental): In total 24 participants will receive two high dose treatments with MV-LASV on day 0 and 28.
  Interventions: Biological: MV-LASV
- Placebo: treatment group C (Placebo Comparator): In total 12 participants will receive placebo treatment on day 0 and 28.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MV-LASV — The MV-LASV vaccine candidate is a recombinant live attenuated viral vectored vaccine, based on the backbone of the measles Schwarz virus strain for prophylaxis of Lassa infection and will be administered in two different dose levels by intra muscular (i.m.) injection.
  Arms: MV-LASV high dose: treatment group B; MV-LASV low dose: treatment group A
Other: Placebo — A sterile physiological saline solution will be used as placebo to ensure blinding of the treatment with low dose MV-LASV and placebo within treatment group A. Additionally, the Placebo will be used as a control arm to enable comparison of treatment reactions within treatment groups B and C.
  Arms: MV-LASV low dose: treatment group A; Placebo: treatment group C

SUMMARY:
This is a randomized, placebo-controlled, single-center, dose finding phase I trial in healthy adult volunteer participants consisting of two phases, an unblinded dose escalation and an observer-blinded treatment phase.

The aim is to investigate the safety, tolerability and immunogenicity of MV-LASV after administration of two different dose levels of MV-LASV. Placebo will be applied to blind the different Treatment schedules.

DETAILED DESCRIPTION:
This is a prospective, interventional, observer-blinded, randomized, phase I trial, comparing different dose levels of MV-LASV. As safety precaution, the study will begin with enrollment of two successive unblinded dose groups of sentinel participants randomized into groups of four in an open-label fashion (group A and B).

Thereafter, 52 participants will be enrolled in an observer-blinded, randomized manner into one of the three treatment groups (A, B or C). Placebo will be applied to blind the different Treatment schedules.

After the screening visit, participants will bei enrolled to one of three Treatment groups. Visits for immunogenicity sample collection and safety assessments will be performed for 56 days, and additionally subjects will for long-term follow-up up to 365 days.

The investigator and site personnel assessing Adverse Events (AEs), all participants, as well as the sponsor's representatives involved in the monitoring and conduct of the study will be unblinded to which vaccine was administered within the unblinded treatment phase. Only the site personnel performing randomization, reparation and administration of Investigational Medicinal Product (IMP) will be unblinded within the randomized observer-blinded treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained before any trial-related activities
2. Healthy men or women aged 18 to ≤ 55 years on the day of consenting
3. Ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to cooperate with the investigator and to comply with the requirements of the entire study
4. All female participants of childbearing potential, defined as all woman physiologically capable of becoming pregnant, must have a negative pregnancy test at screening
5. Willingness not to become pregnant or to father a child during the study up to 182 days after the first vaccination by practicing reliable methods of contraception
6. Availability during the duration of the trial

Exclusion Criteria:

1. Participation in another investigational clinical study (including exposure to an IMP or device) within four weeks before the screening visit or planned concurrent participation in another clinical study before study completion
2. History of immunodeficiency, known HIV infection or current hepatitis B/C infection
3. History of drug addiction including alcohol dependence within the last two years
4. Inability or unwillingness to avoid intake of more than around 20g alcohol per day during 48 hours after each vaccination
5. Vaccination within four weeks prior to first vaccination or planning to receive any non-study vaccine within 182 days after the first vaccination
6. Prior receipt of any Lassa vaccine
7. Recent infection within one week prior to Screening visit
8. Blood donations including plasma donations, 90 days prior to Screening visit and anticipated blood, plasma, tissue, sperm or organ donation, throughout the study until end of treatment period
9. Clinically relevant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, hematological, endocrine, inflammatory, autoimmune or neurological diseases or clinically relevant abnormal laboratory values, that in the opinion of the investigator may interfere with the aim of the study
10. History of neoplastic disease (excluding non-melanoma skin cancer that was successfully treated) within the past five years or a history of any hematological malignancy
11. Behavioral, cognitive, or psychiatric condition that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the study protocol
12. History of severe adverse reactions to vaccine administration, including anaphylaxis and related symptoms, such as urticaria, respiratory difficulty, angioedema and abdominal pain to vaccines, or history of allergic reaction likely to be exacerbated by any component of the vaccine
13. History of or present hearing deficit
14. Present thrombocytopenia and/or history of thrombocytopenia and/or bleeding disorders.
15. History of anaphylaxis to drugs or other allergic reactions, which the investigator considers compromising the safety of the volunteer
16. Use of medication during two weeks before the first vaccination and throughout the study, which the investigator considers affecting the validity of the study, except hormonal contraception or hormonal replacement therapy in female participants (prior to taking any medication within 72 hours before study vaccination, the participant should consult the investigator)
17. Use of immunosuppressive drugs like corticosteroids (excluding topical preparations) within 30 days prior to the first vaccination or anticipated use before completion of day 182
18. Receipt of blood products or immunoglobulins within 120 days prior to the Screening Visit or anticipated receipt of any blood product or immunoglobulin before completion of day 182
19. Pregnancy or lactation at screening or planning to become pregnant before completion of day 182
20. Unreliable contraception Methods
21. Persons in a direct relationship with the sponsor, an investigator or other study team members. Direct dependent relationships include close relatives (i.e. children, parents, partner/spouse, siblings) as well as employees of the clinical study site or the sponsor
22. Individuals who are living and/or working with severely immunocompromised people, children under 15 months old or pregnant women
23. Participants who travelled within one year prior to the first vaccination or plan to travel during the study to an endemic country
24. A rash, dermatological condition or tattoos that would, in the opinion of the Investigator, interfere with injection site reaction rating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Rate of solicited and unsolicited Adverse Events (AEs) | 56 days
  Rate of solicited and unsolicited adverse events (AEs) during the treatment period up to day 56

SECONDARY OUTCOMES:
Rate of Serious Adverse Events (SAEs) | 365 days
  Rate of Serious Adverse Events (SAEs) during the treatment period up to study day 365
Cell-mediated immunity as confirmed by the presence of functional CD4+ and CD8+ T-cells | 56 days
  Cell-mediated immunity specific for LASV up to day 56 as confirmed by the presence of functional CD4+ and CD8+ T-cells
Measurement of anti-LASV antibodies determined by Enzyme-linked Immunosorbent Assay (ELISA) | 56 days
  Measurement of anti-LASV antibodies up to day 56 determined by Enzyme-linked Immunosorbent Assay (ELISA)
Quantification of functional, neutralizing antibodies via Virus Neutralization Tests (VNT) | 56 days
  Quantification of functional, neutralizing antibodies on days 0, 28 and 56 via Virus Neutralization Tests (VNT)
Rate of abnormal laboratory parameters | 56 days
  Rate of abnormal laboratory parameters until day 56
RT-qPCR Analysis of MV-LASV Viral Vector in Human Blood, Urine, and Saliva Samples | 42 days
  Shedding of live recombinant virus up to day 42

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- University of Antwerpen, Centre for the Evaluation of Vaccination (CEV), Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Tschismarov R, Van Damme P, Germain C, De Coster I, Mateo M, Reynard S, Journeaux A, Tomberger Y, Withanage K, Haslwanter D, Terler K, Schrauf S, Mullner M, Tauber E, Ramsauer K, Baize S. Immunogenicity, safety, and tolerability of a recombinant measles-vectored Lassa fever vaccine: a randomised, placebo-controlled, first-in-human trial. Lancet. 2023 Apr 15;401(10384):1267-1276. doi: 10.1016/S0140-6736(23)00048-X. Epub 2023 Mar 16. PMID 36934733